CLINICAL TRIAL: NCT06269276
Title: Caregiver Contribution to Self-Care in Ostomy Patient Index: Turkish Validity and Reliability Study
Status: Completed | Type: Observational
Sponsor: Namik Kemal University (Other)
Responsible Party: Principal Investigator, Tülin YILDIZ, Prof. Dr., Namik Kemal University
Other Study IDs: CAVCU
Record Dates: First submitted 2024-02-12; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Stoma Colostomy; Stoma Ileostomy; Caregiver; Self Care
Keywords: caregiver; stoma; self care

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Caregiver Contribution to Self-Care in Ostomy Patient Index — This study was conducted to evaluate the Turkish validity and reliability of the Caregiver Contribution to Self-Care in Ostomy Patient Index, to evaluate the relatives of patients with stoma who contribute to their self-care in Turkish society, and to contribute to the nursing literature of the measurement tool.

SUMMARY:
This study was conducted to evaluate the Turkish validity and reliability of the Caregiver Contribution to Self-Care in Ostomy Patient Index, to evaluate the relatives of patients with stoma who contribute to their self-care in Turkish society, and to contribute to the nursing literature of the measurement tool.

This methodological type of research was carried out between September 2020 and January 2021 in a state and a university hospital in Tekirdağ. The research sample consisted of 223 individuals who contributed to the self-care of individuals with colostomy, ileostomy and urostomy who applied for outpatient control. In the analysis of the data, descriptive statistics, language and content validity, confirmatory factor analysis, item analysis, internal consistency and test-retest methods were used.

At the end of the study, it was determined that the scale was suitable for Turkish society and was valid and reliable in Turkish.

DETAILED DESCRIPTION:
The "Caregiver Contribution to Self-Care in Ostomy Patient Index" scale consists of 22 items and 3 sub-dimensions. Scale items are evaluated with a 5-point Likert type. The first sub-dimension is "Caregiver Contribution to Self-Care Maintenance" consisting of 9 items; The second sub-dimension is "Caregiver Contribution To Self-Care Monitoring" consisting of 8 items and the third sub-dimension is " Caregiver Contribution to Self-Care Management" consisting of 5 items. The 18th item of the scale, which evaluates the state of experiencing complications, has a low factor load and was accepted as an add-on. The highest 110 points are obtained from the scale, and it is stated that as the total score from the scale increases, self-care also increases.

ELIGIBILITY:
Inclusion Criteria:

* speaking Turkish
* over 18 years old
* Not having a serious psychiatric diagnosis
* Giving written consent to participate in the study

Exclusion Criteria:

* severe visual or auditory problems
* caregivers who did not volunteer to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The research sample consisted of 223 individuals who contributed to the self-care of individuals with colostomy, ileostomy and urostomy who applied for outpatient control.
Sampling Method: Non-Probability Sample
Enrollment: 223 (Actual)
Dates: Start 2020-09-20 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Caregiver Contribution to Self-Care in Ostomy Patient Index | 5 months
  The "Caregiver Contribution to Self-Care in Ostomy Patient Index" scale consists of 22 items and 3 sub-dimensions. Scale items are evaluated with a 5-point Likert type. The first sub-dimension is "Caregiver Contribution to Self-Care Maintenance" consisting of 9 items; The second sub-dimension is "Caregiver Contribution To Self-Care Monitoring" consisting of 8 items and the third sub-dimension is " Caregiver Contribution to Self-Care Management" consisting of 5 items.

CONTACTS AND LOCATIONS:
Locations (1):
- Tekirdag Namık Kemal University, Tekirdağ, Suleymanpasa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided